CLINICAL TRIAL: NCT03909412
Title: Phase I Study of Carfilzomib-based Chemotherapy Mobilization for Autologous Stem Cell Transplantation in Multiple Myeloma
Brief Title: Carfilzomib Based Chemotherapy Mobilization for Autologous Stem Cell Transplants in Multiple Myeloma
Acronym: CarMob
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro2018-0531
Record Dates: First submitted 2019-02-19; First posted 2019-04-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Intervention Model Description: This phase I study utilizes a 3+3 design with escalating cohorts of Carfilzomib at 20mg/m2, 27mg/m2, 36mg/m2, 45mg/m2, 56mg/m2, and 70mg/m2 to be administered concomitantly with Cyclophosphamide 2 gm/m2, Dexamethasone and G-CSF
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Carfilzomib Mobilization - Dose Level 0 (Experimental): Carfilzomib at 20mg/m2 over 10 minutes will be administered concomitantly with Cyclophosphamide 2 gm/m2, Dexamethasone 40mg and G-CSF.
  For patients who are naïve to carfilzomib based therapy a priming dose of Carfilzomib (20mg/m2) will be administered 1 week prior to the cohort dosing.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Granulocyte Colony-Stimulating Factor
- Carfilzomib Mobilization - Dose Level 1 (Experimental): Carfilzomib at 27mg/m2 over 10 minutes will be administered concomitantly with Cyclophosphamide 2 gm/m2, Dexamethasone 40mg and G-CSF.
  For patients who are naïve to carfilzomib based therapy a priming dose of Carfilzomib (20mg/m2) will be administered 1 week prior to the cohort dosing.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Granulocyte Colony-Stimulating Factor
- Carfilzomib Mobilization - Dose Level 2 (Experimental): Carfilzomib at 36mg/m2 over 30 minutes will be administered concomitantly with Cyclophosphamide 2 gm/m2, Dexamethasone 40mg and G-CSF.
  For patients who are naïve to carfilzomib based therapy a priming dose of Carfilzomib (20mg/m2) will be administered 1 week prior to the cohort dosing.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Granulocyte Colony-Stimulating Factor
- Carfilzomib Mobilization - Dose Level 3 (Experimental): Carfilzomib at 45mg/m2 over 30 minutes will be administered concomitantly with Cyclophosphamide 2 gm/m2, Dexamethasone 40mg and G-CSF.
  For patients who are naïve to carfilzomib based therapy a priming dose of Carfilzomib (20mg/m2) will be administered 1 week prior to the cohort dosing.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Granulocyte Colony-Stimulating Factor
- Carfilzomib Mobilization - Dose Level 4 (Experimental): Carfilzomib at 56mg/m2 over 30 minutes will be administered concomitantly with Cyclophosphamide 2 gm/m2, Dexamethasone 40mg and G-CSF.
  For patients who are naïve to carfilzomib based therapy a priming dose of Carfilzomib (20mg/m2) will be administered 1 week prior to the cohort dosing.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Granulocyte Colony-Stimulating Factor
- Carfilzomib Mobilization - Dose Level 5 (Experimental): Carfilzomib at 70mg/m2 over 30 minutes will be administered concomitantly with Cyclophosphamide 2 gm/m2, Dexamethasone 40mg and G-CSF.
  For patients who are naïve to carfilzomib based therapy a priming dose of Carfilzomib (20mg/m2) will be administered 1 week prior to the cohort dosing.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Granulocyte Colony-Stimulating Factor

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib will be administered over 10 minutes for the 20 mg/m2 and 27 mg/m2 dose and over 30 minutes for all higher doses.
  Other Names: Kyprolis
Drug: Cyclophosphamide — Cyclophosphamide dosed at 2gm/m2 administered over 1 hour.
  Other Names: Cytoxan
Drug: Dexamethasone — Dexamethasone 40mg IV/PO to be administered as a premedication.
  Other Names: Decadron
Drug: Granulocyte Colony-Stimulating Factor — On day 7 subjects will initiate high dose G-CSF injections at 14mcg/kg daily (with a cap of 1440mcg daily).
  Other Names: G-CSF; Filgrastim; Neupogen

SUMMARY:
This phase I study utilizes a 3+3 design with escalating cohorts of Carfilzomib at 20mg/m2, 27mg/m2, 36mg/m2, 45mg/m2, 56mg/m2, and 70mg/m2 to be administered concomitantly with Cyclophosphamide 2 gm/m2, Dexamethasone and Granulocyte colony-stimulating factor (G-CSF)

DETAILED DESCRIPTION:
This study will be conducted as an open-label Phase I, single-center study in which subjects will receive carfilzomib, in combination cyclophosphamide and dexamethasone, for mobilization of peripheral blood stem cells. Study treatment will be administered in sequential cohorts, with three to six subjects in each cohort.

Following induction therapy, eligible patients will complete screening procedures. Treatment will consist of Dexamethasone 40mg IV/PO to be administered as a premedication. Carfilzomib dosed at each respective cohort level to be administered over 30 minutes followed by Cyclophosphamide dosed at 2gm/m2 administered over 1 hour.

For patients who are naïve to carfilzomib based therapy a priming dose of Carfilzomib (20mg/m2) will be administered 1 week prior to the cohort dosing.

On day 7 subjects will initiate high dose G-CSF injections at 14mcg/kg daily (with a cap of 1440mcg daily). On day 12 peripheral blood stem cell collection will begin per institutional protocol.

After successful peripheral blood stem cell mobilization, patients will proceed to a melphalan based autologous stem cell transplant.

Patients will have disease parameters assessed monthly after the transplant.

ELIGIBILITY:
INCLUSION CRITERIA Subject has voluntarily agreed to participate by giving written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care. Informed Consent must be obtained prior to mobilization.

* Subject has a confirmed diagnosis of multiple myeloma as specified by the International Myeloma Working Group criteria and must have measurable disease as defined by at least one of the following criteria:
* Serum monoclonal protein ≥ 0.5 g/dL
* ≥200 mg of monoclonal protein in the urine on 24-hour electrophoresis
* Serum immunoglobulin free light chain: involved FLC ≥ 10 mg/dL (≥ 100 mg/L) AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* MRD positivity in peripheral blood by flow cytometry.
* Subject previously received treatment with Carfilzomib.
* Subject is ≥18 years of age at the time of signing the informed consent form.
* Subject has an ECOG performance status of < 2.
* Subjects must have completed any "induction therapy" and have achieved less than a CR.
* Subject has a life expectancy of >12 weeks.

  * Absolute neutrophil count (ANC) ≥1000 cells/mm3 (≥500 for patients with bone marrow biopsy displaying >50% involvement by myeloma)
  * Platelets count ≥ 50,000/mm3 (≥ 30,000 for patients with bone marrow biopsy displaying >50% involvement by myeloma)
  * Hemoglobin > 9.0 g/dL
  * Serum SGOT/AST <3.0 x upper limits of normal (ULN)
  * Serum SGPT/ALT <3.0 x upper limits of normal (ULN)
  * Serum total bilirubin <1.5 x ULN
* Subject must have a MUGA scan or echo with LVEF ≥40% within 6 months of enrollment.
* Females of childbearing potential (FCBP) must have a negative serum pregnancy test should be done within 7 days of treatment initiation and a negative urine pregnancy test within the 24 hours prior to the first study drug administration
* FCBP and male subjects who are sexually active with FCBP must agree to use 2 highly effective concomitant methods of contraception including a male condom during the study and for 90 days following the last dose of study treatment
* Male subjects must agree to not donate sperm while taking carfilzomib and for 90 days after the last dose of carfilzomib.

EXCLUSION CRITERIA

* Subject has a history of allergic reactions to compounds containing captisol, or Carfilzomib
* Subject has a NYHA Class III or IV heart disease and/or a history of active unstable angina, congestive heart disease, severe uncontrolled cardiac arrhythmia, electrocardiographic evidence of acute ischemia, active conduction system abnormalities or myocardial infarction within 6 months prior to enrollment. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
* Uncontrolled hypertension.
* Pulmonary hypertension.
* Known HIV infection, hepatitis C infection (subjects with hepatitis C that achieve a sustained virologic response after antiviral therapy are allowed), or hepatitis B infection (subjects with hepatitis B surface antigen or core antibody that achieve sustained virologic response with antiviral therapy are permitted with a requirement for regular monitoring for reactivation for the duration of treatment on the study).
* Subject has active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Subject has concurrent, uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place him/her at unacceptable risk, including, but not limited to, uncontrolled hypertension, uncontrolled diabetes, active uncontrolled infection, and/or acute chronic liver disease (i.e., hepatitis, cirrhosis).
* Subject has ≥Grade 2 peripheral neuropathy.
* Subject has been diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Subject has received radiation therapy within 3 weeks of enrollment. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
* Subject has had prior mobilization or stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 24 Months
  Safety and tolerability will be assessed by clinical review of all relevant parameters including Adverse Events (CTCAE v4.0)
Maximum tolerated dose (MTD) | 28 Days
  To determine the maximum tolerated dose (MTD) of carfilzomib in combination with cyclophosphamide, dexamethasone and G-CSF in mobilizing and collecting peripheral blood stem cells

CONTACTS AND LOCATIONS:
Locations (1):
- Hackensack Meridian Health - John Theurer Cancer Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mark T, Stern J, Furst JR, Jayabalan D, Zafar F, LaRow A, Pearse RN, Harpel J, Shore T, Schuster MW, Leonard JP, Christos PJ, Coleman M, Niesvizky R. Stem cell mobilization with cyclophosphamide overcomes the suppressive effect of lenalidomide therapy on stem cell collection in multiple myeloma. Biol Blood Marrow Transplant. 2008 Jul;14(7):795-8. doi: 10.1016/j.bbmt.2008.04.008. PMID 18541199
- [Background] Bringhen S, Petrucci MT, Larocca A, Conticello C, Rossi D, Magarotto V, Musto P, Boccadifuoco L, Offidani M, Omede P, Gentilini F, Ciccone G, Benevolo G, Genuardi M, Montefusco V, Oliva S, Caravita T, Tacchetti P, Boccadoro M, Sonneveld P, Palumbo A. Carfilzomib, cyclophosphamide, and dexamethasone in patients with newly diagnosed multiple myeloma: a multicenter, phase 2 study. Blood. 2014 Jul 3;124(1):63-9. doi: 10.1182/blood-2014-03-563759. Epub 2014 May 22. PMID 24855212
- [Background] Berenson JR, Hilger JD, Yellin O, Dichmann R, Patel-Donnelly D, Boccia RV, Bessudo A, Stampleman L, Gravenor D, Eshaghian S, Nassir Y, Swift RA, Vescio RA. Replacement of bortezomib with carfilzomib for multiple myeloma patients progressing from bortezomib combination therapy. Leukemia. 2014 Jul;28(7):1529-36. doi: 10.1038/leu.2014.27. Epub 2014 Jan 16. PMID 24429497
- [Background] Siegel DS, Martin T, Wang M, Vij R, Jakubowiak AJ, Lonial S, Trudel S, Kukreti V, Bahlis N, Alsina M, Chanan-Khan A, Buadi F, Reu FJ, Somlo G, Zonder J, Song K, Stewart AK, Stadtmauer E, Kunkel L, Wear S, Wong AF, Orlowski RZ, Jagannath S. A phase 2 study of single-agent carfilzomib (PX-171-003-A1) in patients with relapsed and refractory multiple myeloma. Blood. 2012 Oct 4;120(14):2817-25. doi: 10.1182/blood-2012-05-425934. Epub 2012 Jul 25. PMID 22833546
- [Background] Munshi NC, Tricot G, Barlogie B: Plasma cell neoplasms, in De Vita VT, Hellman S, Rosenberg SA (ed): Cancer : Principles & Practice on Oncology, 6th edition, Philadelphia, PA. Lippincott Williams & Wilkins, 2001, pp 2465-2499
- [Background] Riedel DA, Pottern LM. The epidemiology of multiple myeloma. Hematol Oncol Clin North Am. 1992 Apr;6(2):225-47. PMID 1582971
- [Background] Chang H, Sloan S, Li D, Zhuang L, Yi QL, Chen CI, Reece D, Chun K, Keith Stewart A. The t(4;14) is associated with poor prognosis in myeloma patients undergoing autologous stem cell transplant. Br J Haematol. 2004 Apr;125(1):64-8. doi: 10.1111/j.1365-2141.2004.04867.x. PMID 15015970
- [Background] Kumar S, Giralt S, Stadtmauer EA, Harousseau JL, Palumbo A, Bensinger W, Comenzo RL, Lentzsch S, Munshi N, Niesvizky R, San Miguel J, Ludwig H, Bergsagel L, Blade J, Lonial S, Anderson KC, Tosi P, Sonneveld P, Sezer O, Vesole D, Cavo M, Einsele H, Richardson PG, Durie BG, Rajkumar SV; International Myeloma Working Group. Mobilization in myeloma revisited: IMWG consensus perspectives on stem cell collection following initial therapy with thalidomide-, lenalidomide-, or bortezomib-containing regimens. Blood. 2009 Aug 27;114(9):1729-35. doi: 10.1182/blood-2009-04-205013. Epub 2009 Jun 26. PMID 19561323
- [Background] Giralt S, Stadtmauer EA, Harousseau JL, Palumbo A, Bensinger W, Comenzo RL, Kumar S, Munshi NC, Dispenzieri A, Kyle R, Merlini G, San Miguel J, Ludwig H, Hajek R, Jagannath S, Blade J, Lonial S, Dimopoulos MA, Einsele H, Barlogie B, Anderson KC, Gertz M, Attal M, Tosi P, Sonneveld P, Boccadoro M, Morgan G, Sezer O, Mateos MV, Cavo M, Joshua D, Turesson I, Chen W, Shimizu K, Powles R, Richardson PG, Niesvizky R, Rajkumar SV, Durie BG; IMWG. International myeloma working group (IMWG) consensus statement and guidelines regarding the current status of stem cell collection and high-dose therapy for multiple myeloma and the role of plerixafor (AMD 3100). Leukemia. 2009 Oct;23(10):1904-12. doi: 10.1038/leu.2009.127. Epub 2009 Jun 25. PMID 19554029
- [Background] Giralt S, Vesole DH, Somlo G, Krishnan A, Stadtmauer E, Mccarthy P, Pasquini MC; Blood and Marrow Transplant Clinical Trials Network Multiple Myeloma Working Group. Re: Tandem vs single autologous hematopoietic cell transplantation for the treatment of multiple myeloma: a systematic review and meta-analysis. J Natl Cancer Inst. 2009 Jul 1;101(13):964; author reply 966-7. doi: 10.1093/jnci/djp126. Epub 2009 Jun 17. No abstract available. PMID 19535777
- [Background] Niesvizky R, Siegel D, Michaeli J. Biology and treatment of multiple myeloma. Blood Rev. 1993 Mar;7(1):24-33. doi: 10.1016/0268-960x(93)90021-u. PMID 8467229
- [Background] Mark T, Niesvizky R, Coleman M. Novel agents in myeloma: an exciting saga. Cancer. 2009 Jan 15;115(2):236-42. doi: 10.1002/cncr.24040. No abstract available. PMID 19025986
- [Background] Niesvizky R, Siegel D, Glassman J, Straus D, Fine J, Lyons L, Michaeli J. Impact of early response to sequential high-dose chemotherapy on outcome of patients with advanced myeloma and poor prognostic features. Leuk Lymphoma. 2002 Mar;43(3):607-12. doi: 10.1080/10428190210324. PMID 12002766
- [Background] Niesvizky R, Choy CG, Fine J, Glassman J, Reich L, Straus D, Zhu A, Michaeli J: Impact of initial response on disease progression following tandem peripheral blood stem cell transplants in patients with poor prognosis multiple myeloma. ASH December, 1998. Abstract # 2728.
- [Background] Mazumder A, Kaufman J, Niesvizky R, Lonial S, Vesole D, Jagannath S. Effect of lenalidomide therapy on mobilization of peripheral blood stem cells in previously untreated multiple myeloma patients. Leukemia. 2008 Jun;22(6):1280-1; author reply 1281-2. doi: 10.1038/sj.leu.2405035. Epub 2007 Nov 22. No abstract available. PMID 18033320
- [Background] Demo SD, Buchholz TJ, Laidig GL, Parlati F, Shenk KD, Smyth MS, et al. Biochemical and cellular characterization of the novel proteasome inhibitor PR-171. Blood 2005;106:455a, Abstract 1588.
- [Background] Velcade® (bortezomib) [full prescribing information]. Cambridge, MA: Millennium Pharmaceuticals, Inc.; 2008.
- [Background] Ivancsits D, Nimmanapali R, Sun M, Shenk K, Demo SD, Bennett MK, et al. The proteasome inhibitor PR-171 inhibits cell growth, induces apoptosis, and overcomes de novo and acquired drug resistance in human multiple myeloma cells. Blood 2006;106:452a.
- [Background] Kuhn DJ, Chen Q, Voorhees PM, Strader JS, Shenk KD, Sun CM, Demo SD, Bennett MK, van Leeuwen FW, Chanan-Khan AA, Orlowski RZ. Potent activity of carfilzomib, a novel, irreversible inhibitor of the ubiquitin-proteasome pathway, against preclinical models of multiple myeloma. Blood. 2007 Nov 1;110(9):3281-90. doi: 10.1182/blood-2007-01-065888. Epub 2007 Jun 25. PMID 17591945
- [Background] Mikhael JR, Reeder CB, Libby EN, Costa LJ, Bergsagel PL, Buadi F, Mayo A, Nagi Reddy SK, Gano K, Dueck AC, Stewart AK. Phase Ib/II trial of CYKLONE (cyclophosphamide, carfilzomib, thalidomide and dexamethasone) for newly diagnosed myeloma. Br J Haematol. 2015 Apr;169(2):219-27. doi: 10.1111/bjh.13296. Epub 2015 Feb 13. PMID 25683772
- [Background] Herve Avet-Loiseau eta al., Evaluation of Minimal Residual Disease (MRD) By Next Generation Sequencing (NGS) Is Highly Predictive of Progression Free Survival in the IFM/DFCI 2009 Trial. ASH annual meeting abstracts. Blood 2015 126:191
- [Background] Martinez-Lopez J, Lahuerta JJ, Pepin F, Gonzalez M, Barrio S, Ayala R, Puig N, Montalban MA, Paiva B, Weng L, Jimenez C, Sopena M, Moorhead M, Cedena T, Rapado I, Mateos MV, Rosinol L, Oriol A, Blanchard MJ, Martinez R, Blade J, San Miguel J, Faham M, Garcia-Sanz R. Prognostic value of deep sequencing method for minimal residual disease detection in multiple myeloma. Blood. 2014 May 15;123(20):3073-9. doi: 10.1182/blood-2014-01-550020. Epub 2014 Mar 19. PMID 24646471
- [Background] Rawstron AC, Orfao A, Beksac M, Bezdickova L, Brooimans RA, Bumbea H, Dalva K, Fuhler G, Gratama J, Hose D, Kovarova L, Lioznov M, Mateo G, Morilla R, Mylin AK, Omede P, Pellat-Deceunynck C, Perez Andres M, Petrucci M, Ruggeri M, Rymkiewicz G, Schmitz A, Schreder M, Seynaeve C, Spacek M, de Tute RM, Van Valckenborgh E, Weston-Bell N, Owen RG, San Miguel JF, Sonneveld P, Johnsen HE; European Myeloma Network. Report of the European Myeloma Network on multiparametric flow cytometry in multiple myeloma and related disorders. Haematologica. 2008 Mar;93(3):431-8. doi: 10.3324/haematol.11080. Epub 2008 Feb 11. PMID 18268286
- [Background] Faham M, Zheng J, Moorhead M, Carlton VE, Stow P, Coustan-Smith E, Pui CH, Campana D. Deep-sequencing approach for minimal residual disease detection in acute lymphoblastic leukemia. Blood. 2012 Dec 20;120(26):5173-80. doi: 10.1182/blood-2012-07-444042. Epub 2012 Oct 16. PMID 23074282